Study Title: The Effects of Exercise Training on Central and Peripheral Blood Flow Regulation in Individuals with Down Syndrome

**Clinical Trial identifier number: NCT04854122** 

**Document date: 03/02/2022** 



### INFORMED CONSENT

# **Department of Physical Therapy**

TITLE OF STUDY: The Effects of Exercise Training on Central and Peripheral Blood Flow

# **Regulation in Individuals With Down Syndrome**

**INVESTIGATOR(S):** Thessa Hilgenkamp

For questions or concerns about the study, you may contact Thessa Hilgenkamp at 702-895-1055.

For questions regarding the rights of research subjects, any complaints or comments regarding the manner in which the study is being conducted, contact the UNLV Office of Research Integrity – Human Subjects at 702-895-2794, toll free at 888-581-2794 or via email at IRB@unlv.edu.

### **Purpose of the Study**

You are invited to participate in a research study. The purpose of this study is to evaluate the effects of an exercise program on regulation of blood pressure, blood flow, gait and balance, and level of support and quality of life in individuals with Down syndrome, compared to a control group without Down syndrome.

### **Participants**

You are being asked to participate in the study because you fit the following criteria:

- You are between 18 and 35 years old
- You are generally healthy
- You have a low active or sedentary lifestyle

#### **Procedures**

If you volunteer to participate in this study, you will be asked to visit a laboratory (the Cardiovascular Research and Exercise Laboratory) on UNLV Campus two times.

During the visits to the laboratory on UNLV Campus, we will start by non-invasively examine cardiac output (how much blood your heart can pump each minute) during a treadmill test. In addition, this study will examine the autonomic response (how your body controls heart rate and blood pressure) and how blood vessels change during and after stimulation (handgrip exercise and lower body negative pressure [LBNP – this is where a small vacuum will be created around your legs]).

# Preparation for all visits

TITLE OF STUDY: The Effects of Exercise Training on Central and Peripheral Blood Flow Regulation in Individuals With Down Syndrome

Twenty-four hours prior to each visit, you cannot participate in any exercise, and you are asked to not drink or eat anything with caffeine, or drink alcohol. You cannot eat anything 3 hours before the visit. If you do not refrain from these things prior to the visits, you will be asked to come back another day. Please wear comfortable clothes to exercise in at each visit. UNLV and the CARE-Lab follow state-issued COVID-10 guidelines with regards to face coverings and social distancing.

#### Visit #1

During the first visit, the researcher will review this consent form with you and answer any questions that you may have. If you agree to participate, you will be asked to sign this informed consent form.

If you agree, we will proceed with the study visit as follows:

We will ask some questions about your health, your physical activity level, any fear of falling and level of support and quality of life. You will also perform a few cognitive tests on an iPad. If you are a female, we will need to test your urine to see if you are pregnant. If you are pregnant, you will not be able to participate in this study. We will also measure around your waist and hip, and you will lie on a table to assess your body composition (how much fat, muscle, bone and tissue is in your body) with a DEXA (a machine that looks like an x-ray). Next, your heart function will be measured using cardiac ultrasound (a heart scan). This test will allow us to see an image of your heart on a computer screen. This is the same technology used to image babies while still in the womb. Some ultrasound gel (consisting of salt and water) will be placed on your chest. We will then place the ultrasound probe over your heart to help us obtain a clear image. We will measure how well your heart contracts and relaxes. We will also measure how stiff the arteries are by briefly holding a small sensor on the skin of your wrist, arm and neck.

Second, you will perform the treadmill walking test. This test is performed to obtain maximal oxygen consumption (VO<sub>2</sub>peak) (the best measure available for fitness/work capacity) and maximal heart rate. You will wear a mask over your mouth and nose so we can analyze the air you breathe out during the treadmill test. The start of the treadmill test will be at a comfortable speed for 4 minutes. Then, the incline (slope) will be increased to 2.5% (to simulate walking uphill) and you will continue walking at the same speed for the next 2 minutes. Then, the incline is increased to 5% and you will continue walking at the same speed. Then, the incline is increased with 2.5% every 2 minutes until 12.5% (to simulate a very steep hill), while you continue walking at the same speed. After that, the incline will be kept constant, but the speed will be increased with 0.5 mph (miles per hour) every minute until you get tired and/or cannot keep up with the speed anymore. If you can, you may be running in this last part. During this test, cardiac output (the amount of blood leaving your heart per minute) will be measured using ultrasound. We will do this by touching your skin with a pencil-like ultrasound probe (ped-off probe) for 30 seconds at the end of every 2-minute stage.

Lastly, we will measure your gait and your balance with a number of different tests. We will look at the way you stand, the way you walk at different speeds, the way you walk stairs and make turns. Then we will look at how well you can keep your balance in different circumstance, such as reaching, closing your eyes, and standing on a moving platform. We will use a harness to prevent you from falling. At the end of the first visit, all participants will be provided with an Actigraph and instructions to wear this device for 7 days.

# Visit #2

TITLE OF STUDY: The Effects of Exercise Training on Central and Peripheral Blood Flow Regulation in Individuals With Down Syndrome

Upon arriving to the lab, we will have you go to the bathroom before we start study procedures. Before and during the testing protocol in the lower body negative pressure (LBNP) chamber (at the end of the 5 min of resting before we start with the handgrip exercise) a total of approximately 6 tablespoons of blood will be drawn from a vein in your arm using a needle. This blood will be analyzed for cardiovascular, inflammatory and hormonal biomarkers, and we will also investigate the relationship between cardiovascular outcomes of this study and specific genetic variations.

You will then be asked to lie on your back in the LBNP chamber to perform arterial health assessments and handgrip exercise. Three electrode stickers will be put on your upper body to measure your heart rate. We will also attach a Velcro band around your chest to measure how much you breathe. We will attach a finger cuff around your middle finger of your left hand to measure your blood pressure, and an arm cuff on the right arm just for baseline measures. Lastly, a very sensitive pen-shaped microphone is placed on the wrist (radial artery). This microphone measures how stiff your radial artery is. After resting for 10 minutes, we will ask you to squeeze the handgrip as hard as you can to measure your maximal force. Then, you will perform different handgrip protocols:

- 1) Squeeze the handgrip 3 times for a single contraction at 20% of your hardest effort, 3 times for a single contraction at 40% of your hardest effort.
- 2) Perform rhythmic handgrip exercise at 15%, 30%, and 45% of your hardest effort for 5 minutes, with a 5-minute rest in-between

During this time, arm blood flow will be measured with ultrasound. In addition, forearm oxygen saturation will be measured by Near-infrared system on the palm side of the right forearm before and during handgrip exercise. A small near-infrared probe will be attached to your right forearm. Next, the LBNP portion of the test will begin. The LBNP will be turned on to a low negative pressure (-20 mmHg) for 5 minutes. The same rhythmic handgrip exercise described in 2) above will be repeated.

Please wear loose and comfortable clothes and shoes that are suitable for working out.

### **Blood Banking**

We would like to save any blood that is left over after we have completed analyzing it for this research study so that it could be used in future research about cardiovascular disease. Upon completion of the study, any remaining samples will be de-identified so that there is no link to your identity. The samples will be stored indefinitely at UNLV in the freezers located in the Translational Biomarker Unit. These de-identified samples could be used for future research studies or distributed to other investigators for future research studies. If you agree to bank your leftover samples, you may withdraw your consent at any time **before** study completion by contacting Dr. Hilgenkamp at 702-895-1055. You will not be able to withdraw your consent **after** study completion (when the samples are de-identified) because we will not know which samples are yours.

| I agree to allow my blood samples to be kept by Dr. Hilgenkamp in the UNLV Translational |
|---|
| Biomarker Unit for use by other researchers for future research to learn more about how to prevent, |
| detect, or treat cardiovascular disease. |
| Initials . |

| TITLE OF STUDY: The Effects of Exercise Training on Central and Peripheral Blood Flow Regulation in Individuals With Down Syndrome |
|---|
| I do NOT agree to allow my blood samples to be kept by Dr. Hilgenkamp in the UNLV Translational Biomarker Unit for use by other researchers for future research to learn more about how to prevent, detect, or treat cardiovascular disease. Initials |
| ■ I agree to allow my blood samples to be kept by Dr. Hilgenkamp in the UNLV Translational Biomarker Unit for use by other researchers for future research to learn more about how to preven detect, or treat other health problems. Initials |
| ☐ I do NOT agree to allow my blood samples to be kept by Dr. Hilgenkamp in the UNLV Translational Biomarker Unit for use by other researchers for future research to learn more about how to prevent, detect, or treat other health problems. Initials |
| Participating in Future Studies As an optional part of this study, we would like to bank (indefinitely store) your contact information t contact you in the future about participating in other research studies about cardiovascular health and Down syndrome. If you agree, Dr. Hilgenkamp will keep the following information: your name, address, phone number, e-mail address, date of birth, age, race, sex, weight and height, and whether you are a control subject or have Down Syndrome. Access will be limited to her alone. You may withdraw your consent at any time in the future by contacting Dr. Hilgenkamp directly at 702-895-1055. |
| ☐ I agree to allow the researchers to contact me about future research. Initials |
| ☐ I do NOT agree to allow the researchers to contact me about future research. Initials |
| Benefits of Participation |

There may not be direct benefits to you as a participant in this study. However, we hope to learn whether exercise can improve the regulation of blood pressure and blood flow in individuals with Down syndrome, and how we need to use this knowledge in motivating and supporting individuals with Down syndrome in an active lifestyle.

# **Risks of Participation**

There are risks involved in all research studies. We consider this research to have minimal risk for the participants because any harm or discomfort anticipated in the research are not greater than in daily life or during the performance of routine physical examinations or tests in the doctor's office or physical therapist's office.

- 1. You may feel uncomfortable providing personal information in the questionnaires. You will be instructed to skip any questions they do not wish to answer.
- 2. Blood pressure will be measured using a cuff around the finger and around the arm. You may

TITLE OF STUDY: The Effects of Exercise Training on Central and Peripheral Blood Flow Regulation in Individuals With Down Syndrome

feel some tingling on the finger and some squeezing on the arm.

- 3. Skin redness may appear where the electrodes (patches) are placed on the skin for heart rate measurements.
- 4. Aerobic capacity test: The treadmill testing may result in muscle soreness, feeling tired, or out of breath. The soreness should go away in a few days. You may also feel dizzy, faint, trip, fall, or sprain an ankle during the testing. Spotters will be used during the test. A mouthpiece will be worn to measure breathing so participants may feel uncomfortable. You may feel warm during the test. Ambient temperature will be kept at a comfortable temperature between 22-24 degrees Celsius. Additional fans will be provided, as needed, to keep you cool and comfortable. You will be instructed that you can stop the test at any time. Other rare, but serious, risks associated with a peak exercise test include: rapid or irregular heart rhythms, chest pain, heart attack, and very rarely death.
- 5. Adverse events and injuries during the exercise testing might occur. Your physical response of will be monitored throughout the test by trained research staff. There have previously not been any problems with adverse events and injuries when the research is performed by experienced personnel, but, in the instance of an adverse event, the PI will report the event to the IRB.
- 6. Risk of loss of privacy or confidentiality of information. To reduce the risk, all data will be stored coded.
- 7. You may experience mild pain, bleeding or bruising at the site of the blood draw. You may also faint or get a mild infection at the site of the draw.
- 8. You may also feel dizzy or light-headed during the tilt-table testing.
- 9. Your hands may get tired squeezing during the hand grip exercise.
- 10. There are no known risks with ultrasound and all efforts will be made to maintain your modesty. The gel used during the ultrasound may feel cool and sticky and is hypoallergenic (not likely to cause an allergic reaction) and washes off easily.

### **Cost /Compensation**

There will not be any financial cost to you to participate in this study. The study will take 5 hours or your time for the study visits to the laboratory. You will be compensated for your time with \$25 for each of the 2 study visits to the laboratory at UNLV Campus. We will do our very best to prevent any injury from happening to you. However, UNLV may not provide compensation if unanticipated injury occurs during the research.

## **Confidentiality**

All information gathered in this study will be kept as confidential as possible. Participants will be asked to provide their mailing address and date of birth for compensation purposes. These identifiers will not be linked to the study data and destroyed upon the completion of the study. No reference will be made in written or oral materials that could link you to this study. All records will be stored in a locked facility at UNLV for 7 years after completion of the study. After the storage time the information gathered will be destroyed.

### **Voluntary Participation**

Your participation in this study is voluntary. You may refuse to participate in this study or in any part of this study. You may withdraw at any time without prejudice to your relations with UNLV. There is

| TITLE OF STUDY: The Effects of Exercise Training on Central and Peripher | al Blood Flow Regulation in Individuals With Down Syndrome |
|---|---|
| no penalty if you withdraw from this study. You are obeginning or any time during the research study. | encouraged to ask questions about this study at the |
| Participant Consent: I have read the above information and agree to partic questions about the research study. I am at least 18 y to me. | |
| Signature of Participant | Date |
| Participant Name (Please Print) | |
| Signature of Investigator | Date |
| Thessa Hilgenkamp Investigator Name (Please Print) | |